CLINICAL TRIAL: NCT06137703
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, 4-PERIOD, 4-WAY CROSSOVER, RELATIVE BIOAVAILABILITY STUDY OF ZAVEGEPANT (BHV-3500) ORAL FORMULATIONS UNDER FASTING CONDITIONS
Brief Title: A Study to Learn About the Study Medication, Zavegepant, in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BHV3500-113; C5301003 (Other: Alias Study Number)
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-06

CONDITIONS: Biological Availability

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, single dose, 4-period cross-over, comparative bioavailability study in healthy volunteer participants.
Masking Description: All investigators, Sponsor personnel, clinical monitors, independent PK analyst, and participants in the study will be unblinded to the treatment allocation as the primary and secondary endpoints are based on objective criteria of laboratory findings.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (Experimental): Period 1 - Single zavegepant 100mg non-enteric coated soft gel capsule (Treatment A) followed by at least 7 days washout; Period 2 - Two zavegepant 100mg immediate release tablets (Treatment C) followed by at least 7 days washout; Period 3 - Single zavegepant 100mg immediate release tablet (Treatment B) followed by at least 7 days washout; Period 4 - Four zavegepant 25mg enteric coated soft gel capsule (Treatment D).
  Interventions: Drug: Zavegepant 100mg non-enteric coated soft gel capsule; Drug: Zavegepant 100mg immediate release tablet; Drug: Zavegepant 2 x 100mg immediate release tablets; Drug: Zavegepant 4 x 25mg enteric coated soft gel capsule
- Sequence 2 (Experimental): Period 1 - Two zavegepant 100mg immediate release tablets (Treatment C) followed by at least 7 days washout; Period 2 - Four zavegepant 25mg enteric coated soft gel capsule (Treatment D) followed by at least 7 days washout; Period 3 - Single zavegepant 100mg non-enteric coated soft gel capsule (Treatment A) followed by at least 7 days washout; Period 4 - Single zavegepant 100mg immediate release tablet (Treatment B).
  Interventions: Drug: Zavegepant 100mg non-enteric coated soft gel capsule; Drug: Zavegepant 100mg immediate release tablet; Drug: Zavegepant 2 x 100mg immediate release tablets; Drug: Zavegepant 4 x 25mg enteric coated soft gel capsule
- Sequence 3 (Experimental): Period 1 - Single zavegepant 100mg immediate release tablet (Treatment B) followed by at least 7 days washout; Period 2 - Single zavegepant 100mg non-enteric coated soft gel capsule (Treatment A) followed by at least 7 days washout; Period 3 - Four zavegepant 25mg enteric coated soft gel capsule (Treatment D) followed by at least 7 days washout; Period 4 - Two zavegepant 100mg immediate release tablets (Treatment C).
  Interventions: Drug: Zavegepant 100mg non-enteric coated soft gel capsule; Drug: Zavegepant 100mg immediate release tablet; Drug: Zavegepant 2 x 100mg immediate release tablets; Drug: Zavegepant 4 x 25mg enteric coated soft gel capsule
- Sequence 4 (Experimental): Period 1 - Four zavegepant 25mg enteric coated soft gel capsule (Treatment D) followed by at least 7 days washout; Period 2 - Single zavegepant 100mg immediate release tablet (Treatment B) followed by at least 7 days washout; Period 3 - Two zavegepant 100mg immediate release tablets (Treatment C) followed by at least 7 days washout; Period 4 - Single zavegepant 100mg non-enteric coated soft gel capsule (Treatment A).
  Interventions: Drug: Zavegepant 100mg non-enteric coated soft gel capsule; Drug: Zavegepant 100mg immediate release tablet; Drug: Zavegepant 2 x 100mg immediate release tablets; Drug: Zavegepant 4 x 25mg enteric coated soft gel capsule

INTERVENTIONS:
Drug: Zavegepant 100mg non-enteric coated soft gel capsule — Zavegepant (PF-07930207/BHV3500) 100mg non-enteric coated soft gel capsule
  Other Names: Treatment A
Drug: Zavegepant 100mg immediate release tablet — Zavegepant (PF-07930207/BHV3500) 100mg dodecylmaltoside dosage form immediate release tablet
  Other Names: Treatment B
Drug: Zavegepant 2 x 100mg immediate release tablets — 2 x Zavegepant (PF-07930207/BHV3500) 100mg dodecylmaltoside dosage form immediate release tablets - total dose 200mg
  Other Names: Treatment C
Drug: Zavegepant 4 x 25mg enteric coated soft gel capsule — Zavegepant (PF-07930207/BHV3500) 25 mg enteric coated soft gel capsules - total dose 100mg
  Other Names: Treatment D

SUMMARY:
This trial is designed to compare the rate and extent of absorption of four different formulations of zavegepant. 52 healthy male and female volunteers will receive a single dose of each formulation at least 7 days apart over a period of about 7 weeks and the amount of drug in their blood will be assessed over the 24 hour period after each dose.

DETAILED DESCRIPTION:
This is a Phase 1, single centre, open-label, single dose, 4-period, crossover study designed to compare the pharmacokinetics (PK) of zavegepant from three Test products and a Reference product (treatment D).

52 male and female healthy volunteers will be randomly assigned to one of 4 treatment sequences: ACBD, CDAB, BADC, and DBCA.

In each period, subjects will receive one of the following: Treatment A, B, C, or D on Day 1, followed by 24 hours of PK and safety assessments. On Day 2 subjects will be discharged from the clinical site and instructed to return after at least a 7 day washout time has passed for subsequent periods of treatment.

The study will include a screening visit from Day -28 to Day -2. Eligible subjects will be admitted to the clinical site on Day -1 and will be confined until completion of the assessments on Day 2. There will be a washout period of at least 7 days between doses. Study Exit procedures will be performed after the last assessment on the morning of Day 2 of Period 4. Study Exit procedures will be performed as soon as possible in case of Early Termination.

The total duration of study participation for each subject from Screening through Study Exit is anticipated to be approximately 6.5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants must provide Informed Consent Form (ICF) obtained prior to the conduct of any study activities.
* Healthy Male or female participants at least 18 and less than 56 years of age,
* Participants must be Non-smokers and not have used any nicotine-containing products for 3 months prior to screening.
* Body Mass Index (BMI) >18.5 and <30.0kg/m2 and body weight ≥ 50.0kg for males and ≥ 45.0kg for females.
* All females participants must not be breastfeeding and have a negative urine pregnancy test at Screening.
* Females of childbearing potential must be willing to use acceptable contraceptive methods throughout the study and for 30 days after the last study drug administration.
* Male participants with a female partner of childbearing potential must be willing to use acceptable contraceptive methods from the first study drug administration until at least 90 days after the last study drug administration.

Exclusion Criteria:

* Current diagnosis of viral hepatitis or a history of liver disease.
* Any history of seizure disorder (e.g., epilepsy) other than a single childhood febrile seizure.
* Current or recent (within 3 months of the first study drug administration) gastrointestinal disease that may interfere with drug absorption.
* Prior gastrointestinal surgery that interferes with absorption and motility (e.g., gastric bypass, duodenectomy or gastric banding).
* History of drug or alcohol abuse.
* History of anaphylaxis, a documented hypersensitivity reaction, or a clinically significant reaction to any drug or to any of the excipient supporting the zavegepant formulations.
* Donation of plasma within 7 days prior to dosing, or donation or loss of blood (excluding volume drawn at Screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to dosing.
* Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the dosing, extended to 90 days for biological products.
* Inability or difficulty to swallow tablets or capsules.
* Subjects with any clinically significant abnormality or significant abnormal laboratory test results found during medical screening or Day-1. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody during screening.
* Inadequate renal function - estimated glomerular filtration rate (eGFR) according to the Modification of Diet in Renal Disease (MDRD) study equation ≤ 60 mL/min/1.73 m2 at Screening.
* Any of the following laboratory parameters greater than the upper limit of normal (ULN) values at Screening or Baseline (Day -1): alkaline phosphatase (ALP) aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, direct bilirubin, and indirect bilirubin, and alkaline phosphatase.
* Any clinically significant abnormalities on 12-lead ECG or blood pressure (BP) at Screening or Baseline (Day -1) visits.
* Any clinically significant abnormal haematological laboratory test values at Screening or Baseline (Day -1) visits.
* Positive test for COVID-19 performed on Day -1 of each period.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Syneos Health Clinical Research Services, Llc, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=BHV3500-113

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 52 participants were assigned to study interventions.
Groups:
- Sequence DBCA: Participants were assigned to Sequence DBCA, and received a single dose of study intervention on Day 1 of each period per the sequence. There was a washout period of at least 7 days between doses. A=1×100-mg zavegepant non-enteric coated soft gelatin capsule (SGC) administered under fasting condition. B=1×100-mg zavegepant immediate release (IR) tablet + dodecylmaltoside (DDM) dosage form administered under fasting condition. C=1×200-mg zavegepant IR tablet (total dose of 200 mg) + DDM dosage form administered under fasting condition. D=4×25-mg zavegepant enteric coated SGC (total dose of 100 mg) administered under fasting condition.
- Sequence BADC: Participants were assigned to Sequence BADC, and received a single dose of study intervention on Day 1 of each period per the sequence. There was a washout period of at least 7 days between doses. A=1×100-mg zavegepant non-enteric coated SGC administered under fasting condition. B=1×100-mg zavegepant IR tablet + DDM dosage form administered under fasting condition. C=1×200-mg zavegepant IR tablet (total dose of 200 mg) + DDM dosage form administered under fasting condition. D=4×25-mg zavegepant enteric coated SGC (total dose of 100 mg) administered under fasting condition.
- Sequence ACBD: Participants were assigned to Sequence ACBD, and received a single dose of study intervention on Day 1 of each period per the sequence. There was a washout period of at least 7 days between doses. A=1×100-mg zavegepant non-enteric coated SGC administered under fasting condition. B=1×100-mg zavegepant IR tablet + DDM dosage form administered under fasting condition. C=1×200-mg zavegepant IR tablet (total dose of 200 mg) + DDM dosage form administered under fasting condition. D=4×25-mg zavegepant enteric coated SGC (total dose of 100 mg) administered under fasting condition.
- Sequence CDAB: Participants were assigned to Sequence CDAB, and received a single dose of study intervention on Day 1 of each period per the sequence. There was a washout period of at least 7 days between doses. A=1×100-mg zavegepant non-enteric coated SGC administered under fasting condition. B=1×100-mg zavegepant IR tablet + DDM dosage form administered under fasting condition. C=1×200-mg zavegepant IR tablet (total dose of 200 mg) + DDM dosage form administered under fasting condition. D=4×25-mg zavegepant enteric coated SGC (total dose of 100 mg) administered under fasting condition.
Period: Overall Study
Arm/Group | Sequence DBCA | Sequence BADC | Sequence ACBD | Sequence CDAB
Started | 13 | 13 | 13 | 13
Completed | 13 | 12 | 12 | 13
Not Completed | 0 | 1 | 1 | 0
Not completed — Other | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Included all participants who received at least 1 dose of any study intervention.
Groups:
- All Participants: Participants were assigned to 1 of the 4 sequences, and each sequence consisted of 4 periods. The 4 sequences were ACBD, CDAB, BADC, and DBCA. There was a washout period of at least 7 days between doses. A=1×100-mg zavegepant non-enteric coated SGC administered under fasting condition. B=1×100-mg zavegepant IR tablet + DDM dosage form administered under fasting condition. C=1×200-mg zavegepant IR tablet (total dose of 200 mg) + DDM dosage form administered under fasting condition. D=4×25-mg zavegepant enteric coated SGC (total dose of 100 mg) administered under fasting condition.
Arm/Group | All Participants
Number analyzed (Participants) | 52
Age, Customized [Median (Full Range); unit: Years]
  18-65 years of age | 37.0 [22 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 51
  Not Hispanic or Latino | 1
  Not Reported | 0
  Unknown | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian | 0
  Asian | 0
  Black | 11
  Hawaiian | 0
  White | 41
  Multiple | 0
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) of Zavegepant
Description: AUCinf was calculated as AUClast+(Clast*/kel), where AUClast is the area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration, Clast* is the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis, and kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. AUClast was calculated using Linear/Log trapezoidal method.
Time Frame: Pre-dose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16, and 24 hours post dose
Population: Included all participants who received at least 1 dose of zavegepant, and for whom the pharmacokinetic (PK) profile had been adequately characterized.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter (h*ng/mL)
Groups:
- Treatment A: Zavegepant 100 mg SGC: Participants received a single dose of one 100-mg zavegepant non-enteric coated SGC administered under fasting condition on Day 1 of the period assigned.
- Treatment B: Zavegepant 100 mg IR+DDM: Participants received a single dose of one 100-mg zavegepant IR tablet + DDM dosage form under fasting condition on Day 1 of the period assigned.
- Treatment C: Zavegepant 200 mg IR+DDM: Participants received a single dose of one 200-mg zavegepant IR tablet + DDM dosage form administered under fasting condition on Day 1 of the period assigned.
- Treatment D: Zavegepant 4*25 mg SGC: Participants received a single dose of four 25-mg zavegepant (total dose of 100 mg) enteric coated SGCs administered under fasting condition on Day 1 of the period assigned.
Arm/Group | Treatment A: Zavegepant 100 mg SGC | Treatment B: Zavegepant 100 mg IR+DDM | Treatment C: Zavegepant 200 mg IR+DDM | Treatment D: Zavegepant 4*25 mg SGC
Number analyzed (Participants) | 48 | 47 | 47 | 40
Hours*nanograms per milliliter (h*ng/mL) | 83.65 (52) | 102.5 (66) | 184.4 (73) | 47.29 (51)

2. Primary Outcome: Maximum Observed Concentration (Cmax) of Zavegepant
Description: Cmax was observed directly from data.
Time Frame: Pre-dose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16, and 24 hours post dose
Population: Included all participants who received at least 1 dose of zavegepant, and for whom the PK profile had been adequately characterized.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Treatment A: Zavegepant 100 mg SGC: Participants received a signle dose of one 100-mg zavegepant non-enteric coated SGC administered under fasting condition on Day 1 of the period assigned.
Arm/Group | Treatment A: Zavegepant 100 mg SGC | Treatment B: Zavegepant 100 mg IR+DDM | Treatment C: Zavegepant 200 mg IR+DDM | Treatment D: Zavegepant 4*25 mg SGC
Number analyzed (Participants) | 50 | 51 | 50 | 50
ng/mL | 36.28 (68) | 41.20 (80) | 76.93 (77) | 12.78 (82)

3. Primary Outcome: AUClast of Zavegepant
Description: AUClast was calculated using linear/log trapezoidal method.
Time Frame: Pre-dose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16, and 24 hours post dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: Zavegepant 100 mg SGC | Treatment B: Zavegepant 100 mg IR+DDM | Treatment C: Zavegepant 200 mg IR+DDM | Treatment D: Zavegepant 4*25 mg SGC
Number analyzed (Participants) | 50 | 51 | 50 | 50
h*ng/mL | 82.13 (54) | 96.25 (66) | 175.5 (72) | 42.25 (54)

4. Secondary Outcome: Time to Reach Cmax (Tmax) of Zavegepant
Description: Tmax was observed directly from data as time of first occurrence.
Time Frame: Pre-dose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16, and 24 hours post dose
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment A: Zavegepant 100 mg SGC | Treatment B: Zavegepant 100 mg IR+DDM | Treatment C: Zavegepant 200 mg IR+DDM | Treatment D: Zavegepant 4*25 mg SGC
Number analyzed (Participants) | 50 | 51 | 50 | 50
Hours | 0.9830 [0.483 to 3.00] | 0.5000 [0.250 to 2.62] | 0.5000 [0.233 to 2.48] | 2.000 [0.483 to 5.00]

5. Secondary Outcome: Terminal Phase Half-Life (t1/2) of Zavegepant
Description: t1/2 was calculated as Log e(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Pre-dose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16, and 24 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Treatment A: Zavegepant 100 mg SGC | Treatment B: Zavegepant 100 mg IR+DDM | Treatment C: Zavegepant 200 mg IR+DDM | Treatment D: Zavegepant 4*25 mg SGC
Number analyzed (Participants) | 48 | 47 | 47 | 40
Hours | 8.346 (1.3101) | 8.907 (2.3611) | 8.243 (1.3004) | 9.149 (1.5552)

6. Secondary Outcome: Apparent Clearance (CL/F) of Zavegepant From Plasma
Description: CL/F was calculated as dose/AUCinf. AUCinf was calucalted as AUClast+(Clast*/kel), where Clast* is the predicted plasma concentration at the last quantifiable time point estimated, and kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. AUClast was calculated using linear/log trapezoidal method.
Time Frame: Pre-dose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16, and 24 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour (L/h)
Arm/Group | Treatment A: Zavegepant 100 mg SGC | Treatment B: Zavegepant 100 mg IR+DDM | Treatment C: Zavegepant 200 mg IR+DDM | Treatment D: Zavegepant 4*25 mg SGC
Number analyzed (Participants) | 48 | 47 | 47 | 40
liters per hour (L/h) | 1195 (52) | 975.5 (66) | 1085 (73) | 2115 (51)

7. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Zavegepant
Description: Vz/F was calculated by Dose/(AUCinf×kel). AUCinf was calculated by AUClast+(Clast*/kel), where Clast* is the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis, and kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. AUClast was calculated using the linear/log trapezoidal method.
Time Frame: Pre-dose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16, and 24 hours post dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Treatment A: Zavegepant 100 mg SGC | Treatment B: Zavegepant 100 mg IR+DDM | Treatment C: Zavegepant 200 mg IR+DDM | Treatment D: Zavegepant 4*25 mg SGC
Number analyzed (Participants) | 48 | 47 | 47 | 40
L | 14230 (60) | 12250 (79) | 12740 (85) | 27530 (59)

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Adverse evetn (AE)=any untoward medical occurrence in a patient or clinical trial participant administered a pharmaceutical product and which does not necessarily have a causal relationship with the treatment. TEAEs=AEs between first dose of study treatment and up to the end of study participation that were absent before treatment or that worsened relative to pretreatment state. A serious TEAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. SAEs were adjudicated according to the investigator's assessment. Treatment-related was classified based on medical judgement. Severe=Incapacitating with inability to carry out usual activities or significantly affects clinical status, and requires specific action and/or medical attention.
Time Frame: Baseline up to study exit (approximately 6.5 weeks)
Population: Included all participants who received at least 1 dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Zavegepant 100 mg SGC | Treatment B: Zavegepant 100 mg IR+DDM | Treatment C: Zavegepant 200 mg IR+DDM | Treatment D: Zavegepant 4*25 mg SGC
Number analyzed (Participants) | 51 | 51 | 50 | 50
Participants
  Participants with at least 1 TEAE | 3 | 2 | 4 | 3
  Participants with at least 1 treatment-related TEAE | 1 | 0 | 1 | 0
  Participants with at least 1 Severe TEAEs | 1 | 0 | 0 | 1
  Participants with at least 1 Serious TEAEs | 1 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Clinically significant laboratory abnormalities were identified as Grade 3 to 4 laboratory test results graded according to numeric laboratory test criteria in the latest version of Common Technical Criteria for Adverse Events (CTCAE) if available, otherwise according to the latest version of Division of Acquired Immunodeficiency Syndrome (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version. Clinically significant laboratory abnormalities with occurrence in at least 1 participant are reported for this outcome measure. Baseline was defined as the last results (scheduled or unscheduled) obtained prior to the first drug administration.
Time Frame: Baseline up to study exit (approximately 6.5 weeks)
Population: Included all participants who received at least 1 dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Zavegepant 100 mg SGC | Treatment B: Zavegepant 100 mg IR+DDM | Treatment C: Zavegepant 200 mg IR+DDM | Treatment D: Zavegepant 4*25 mg SGC
Number analyzed (Participants) | 52 | 52 | 52 | 52
Participants
  Hematology - Hemoglobin<lower limit of normal | 1 | 0 | 1 | 0
  Urinalysis - Abnormal Leukocyte Esterase | 0 | 0 | 0 | 1
  Urinalysis - Abnormal Urine Leukocytes | 0 | 0 | 0 | 1

10. Secondary Outcome: Blood Pressure on Day -1 and Day 1 of Each Period
Description: Blood pressure was measured after the participants had been resting for at least 5 minutes in a seated position. Normal range for systolic blood pressure (SBP)=90-140 mm Hg; normal range for diastolic blood pressure (DBP)=50-90 mm Hg.
Time Frame: Day -1, pre-dose and 2 hours post dose on Day 1 of each period
Population: Safety analysis set included all participants who received at least 1 dose of any study intervention. Number of Participants Analyzed represents the total number of participants in the safety analysis set. Number Analyzed in each row represents the number of participants with observations at each time point.
Measure: Median (Full Range); unit: millimeter of mercury (mm Hg)
Arm/Group | Treatment A: Zavegepant 100 mg SGC | Treatment B: Zavegepant 100 mg IR+DDM | Treatment C: Zavegepant 200 mg IR+DDM | Treatment D: Zavegepant 4*25 mg SGC
Number analyzed (Participants) | 51 | 51 | 50 | 50
millimeter of mercury (mm Hg)
  SBP on Day -1 | 115.0 [99 to 137] | 115.0 [99 to 140] | 116.5 [94 to 140] | 116.5 [97 to 138]
  Pre-dose SBP on Day 1 of each period | 113.0 [74 to 132] | 113.0 [93 to 132] | 114.0 [92 to 144] | 114.5 [94 to 138]
  SBP at 2 hours post dose on Day 1 of each period | 113.0 [94 to 150] | 114.0 [94 to 135] | 113.5 [91 to 144] | 113.0 [92 to 137]
  DBP at Day -1 | 75.0 [62 to 90] | 77.0 [59 to 89] | 76.0 [64 to 92] | 76.0 [60 to 92]
  Pre-dose DBP on Day 1 of each period | 75.0 [52 to 92] | 76.0 [63 to 90] | 74.0 [64 to 89] | 76.0 [63 to 90]
  DBP at 2 hours post dose on Day 1 of each period | 75.0 [57 to 100] | 76.0 [62 to 97] | 77.0 [61 to 91] | 75.0 [66 to 88]

11. Secondary Outcome: Blood Pressure at Screening and Study Exit
Description: Blood pressure was measured after the participants had been resting for at least 5 minutes in a seated position. Normal range for SBP=90-140 mm Hg; normal range for DBP=50-90 mm Hg.
Time Frame: Screening and study exit
Population: as for outcome 10
Measure: Median (Full Range); unit: mm Hg
Arm/Group | All Participants
Number analyzed (Participants) | 52
mm Hg
  SBP at Screening | 121.5 [102 to 144]
  SBP at study exit | 114.0 [94 to 137]
  DBP at Screening | 82.0 [65 to 91]
  DBP at study exit | 76.0 [63 to 90]

12. Secondary Outcome: Heart Rate (HR) on Day -1 and Day 1 of Each Period
Description: HR was measured after the participants had been resting for at least 5 minutes in a seated position. Normal range for heart rate=50-100 beats/min.
Time Frame: Day -1, pre-dose and 2 hours post dose on Day 1 of each period
Population: as for outcome 10
Measure: Median (Full Range); unit: Beats per minute (beats/min)
Arm/Group | Treatment A: Zavegepant 100 mg SGC | Treatment B: Zavegepant 100 mg IR+DDM | Treatment C: Zavegepant 200 mg IR+DDM | Treatment D: Zavegepant 4*25 mg SGC
Number analyzed (Participants) | 51 | 51 | 50 | 50
Beats per minute (beats/min)
  HR on Day -1 | 71.0 [50 to 102] | 72.0 [49 to 102] | 73.0 [50 to 99] | 73.0 [56 to 100]
  Pre-dose HR on Day 1 of each period | 73.0 [51 to 93] | 74.0 [47 to 99] | 73.5 [52 to 103] | 73.5 [51 to 110]
  HR at 2 hours post dose on Day 1 of each period | 71.0 [51 to 97] | 70.0 [48 to 90] | 71.0 [48 to 108] | 70.0 [50 to 99]

13. Secondary Outcome: HR at Screening and Study Exit
Description: as for outcome 12
Time Frame: Screening and study exit
Population: as for outcome 10
Measure: Median (Full Range); unit: beats/min
Arm/Group | All Participants
Number analyzed (Participants) | 52
beats/min
  HR at Screening | 65.0 [46 to 93]
  HR at study exit | 74.0 [53 to 100]

14. Secondary Outcome: Respiratory Rate (RR) on Day -1 of Each Period
Description: RR was measured after the participants had been resting for at least 5 minutes in a sitting position. Normal range for RR=8-20 breaths/min.
Time Frame: Day -1 of each period
Population: Safety analysis set included all participants who received at least 1 dose of any study intervention. Number of Participants Analyzed represents the total number of participants in the safety analysis set who had at least 1 observation of RR on Day -1.
Measure: Median (Full Range); unit: Breaths per minute (breaths/min)
Arm/Group | Treatment A: Zavegepant 100 mg SGC | Treatment B: Zavegepant 100 mg IR+DDM | Treatment C: Zavegepant 200 mg IR+DDM | Treatment D: Zavegepant 4*25 mg SGC
Number analyzed (Participants) | 46 | 46 | 45 | 45
Breaths per minute (breaths/min) | 14.0 [12 to 18] | 14.0 [12 to 16] | 14.0 [12 to 18] | 14.0 [12 to 18]

15. Secondary Outcome: RR at Screening and Study Exit
Description: as for outcome 14
Time Frame: Screening and study exit
Population: as for outcome 10
Measure: Median (Full Range); unit: breaths/min
Arm/Group | All Participants
Number analyzed (Participants) | 52
breaths/min
  RR at Screening | 14.0 [12 to 16]
  RR at study exit | 14.0 [12 to 18]

16. Secondary Outcome: Temperature on Day -1 of Each Period
Description: Temperature was measured after the participants had been resting for at least 5 minutes in a seated position. Normal range for temperature=35.8-37.6 ℃.
Time Frame: Day -1 of each period
Population: Safety analysis set included all participants who received at least 1 dose of any study intervention. Number of Participants Analyzed represents the total number of participants in the safety analysis set who had at least 1 observation of temperature on Day -1.
Measure: Median (Full Range); unit: Degree Celsius (℃)
Arm/Group | Treatment A: Zavegepant 100 mg SGC | Treatment B: Zavegepant 100 mg IR+DDM | Treatment C: Zavegepant 200 mg IR+DDM | Treatment D: Zavegepant 4*25 mg SGC
Number analyzed (Participants) | 46 | 46 | 45 | 45
Degree Celsius (℃) | 36.60 [36.1 to 37.6] | 36.40 [35.9 to 37.0] | 36.50 [35.9 to 37.2] | 36.50 [36.1 to 37.4]

17. Secondary Outcome: Temperature at Screening and Study Exit
Description: as for outcome 16
Time Frame: Screening and study exit
Population: Included all participants who received at least 1 dose of any study intervention.
Measure: Median (Full Range); unit: ℃
Arm/Group | All Participants
Number analyzed (Participants) | 52
℃
  Temperature at Screening | 36.40 [35.9 to 36.8]
  Temperature at study exit | 36.60 [35.8 to 37.4]

18. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG)
Description: ECG was measured after the participants had been resting for at least 5 minutes in a seated position.
Time Frame: Screening up to study exit (approximately 6.5 weeks)
Population: Included all participants who received at least 1 dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 52
Participants
  ECG Mean Heart Rate | 0
  PR Interval, Aggregate | 0
  QRS Duration, Aggregate | 0
  QT Interval, Aggregate | 0
  QTc corrected using Bazett's formula (QTcB) Interval, Aggregate | 0
  QTc corrected using Fridericia's formula (QTcF) Interval, Aggregate | 0

ADVERSE EVENTS:
Time Frame: Screening up to study exit (approximately 6.5 weeks)
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Treatment A: Zavegepant 100 mg SGC | Treatment B: Zavegepant 100 mg IR+DDM | Treatment C: Zavegepant 200 mg IR+DDM | Treatment D: Zavegepant 4*25 mg SGC
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/51 | 0/51 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 3/51 | 2/51 | 4/50 | 3/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Zavegepant 100 mg SGC (N=51) | Treatment B: Zavegepant 100 mg IR+DDM (N=51) | Treatment C: Zavegepant 200 mg IR+DDM (N=50) | Treatment D: Zavegepant 4*25 mg SGC (N=50)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Zavegepant 100 mg SGC (N=51) | Treatment B: Zavegepant 100 mg IR+DDM (N=51) | Treatment C: Zavegepant 200 mg IR+DDM (N=50) | Treatment D: Zavegepant 4*25 mg SGC (N=50)
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 1
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/03/NCT06137703/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/03/NCT06137703/SAP_001.pdf